CLINICAL TRIAL: NCT06622798
Title: A Retrospective Study Exploring the Correlation Between HRD Score and PARPi Efficacy Based on Chinese Ovarian Cancer Patients
Brief Title: Exploratory Study on the Correlation Between HRD Score and PARPi Efficacy Based on Chinese Ovarian Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Amoy Diagnostics (Industry)
Responsible Party: Principal Investigator, Jing Li, Associate chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2024-218-01
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Exploring the Correlation of HRD Score Pairs with the Prognosis of Chinese Ovarian Cancer Patients and the Outcome of Maintenance Therapy with PARPi
Keywords: HRD; PARPi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — surgical tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
This study plans to retrospectively include 470 initial surgical specimens from 470 patients with epithelial ovarian, fallopian tube or primary peritoneal cancers who were treated with PARPi maintenance therapy in the hospital from 2018.01 to 2024.01. All patients included would be scored by the proprietary HRD ADx-GSS® algorithm with the detecting results of the three genomic statuses including heterozygous omission (LOH), telomere allelic imbalance (TAI), and large-segment translocation (LST). Finally, the correlation between the HRD scores and the prognosis of Chinese ovarian cancer patients and the efficacy of using PARPi as maintenance treatment would be explored.

DETAILED DESCRIPTION:
Although most advanced ovarian cancers achieve clinical remission after conventional initial treatment, the recurrence rate is still high in clinics. Poly ADP-ribose polymerase inhibitor (PARPi) is widely used in the maintenance treatment of ovarian cancer after chemotherapy to prolong the time to recurrence, and its main mechanism is to inhibit the repair of single-stranded DNA damage in tumour cells, which is synthetically lethal in the tumour cells with mutations in the BRCA1/2 gene. Numerous studies have shown that homologous recombination deficiency (HRD) exists in about 50% of epithelial ovarian cancer patients, and has been confirmed to be a predictor of ovarian cancer patients' response to PARPi therapy. However, up to now, there is still no uniform scoring and threshold standard for HRD detection in China. With the increasing attention of HRD detection in clinical diagnosis and treatment, acknowledged standards of HRD scoring algorithms and thresholds are essential. Using a retrospective. Thus, this observational and retrospective study intends to enroll 470 patients with epithelial ovarian, fallopian tube or primary peritoneal cancers who were treated with PARPi maintenance therapy in the hospital from 2018.01 to 2024.01. All patients included would be scored by the proprietary HRD ADx-GSS® algorithm with the detecting results of the three genomic statuses including heterozygous omission (LOH), telomere allelic imbalance (TAI), and large-segment translocation (LST). Finally, the correlation between the HRD scores and the prognosis of Chinese ovarian cancer patients and the efficacy of using PARPi as maintenance treatment would be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer initially diagnosed after January 2015 or platinum-sensitive recurrent patients diagnosed with advanced epithelial ovarian, fallopian tube, and primary peritoneal cancers, and are treated with PARPi maintenance therapy by January 2024 after chemotherapy or Platinum-sensitive recurrent patients diagnosed with advanced epithelial ovarian, fallopian tube, and primary peritoneal cancers, and are treated with PARPi maintenance therapy by January 2024 after chemotherapy;
2. Age ≥ 18 years, female;
3. Stable CA125 level, ECOG: 0-2 points, and appropriate cardiac, liver and renal function before using PARPi.

Exclusion Criteria:

1. other malignancies combined within 5 years;
2. poor underlying condition, one of the following: ECOG PS score >2, KPS score <60, cardiac insufficiency (Class III-IV), hepatic insufficiency (Child-Pugh Class C), renal insufficiency (Stage 4-5);
3. patients whose sample residuals and quality do not support the need for testing;
4. conditions that, in the judgement of the investigator, may affect the conduct of the clinical study and the determination of the study results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study was conducted in female patients with advanced epithelial ovarian, fallopian tube, and primary peritoneal cancers
Study Population: Patients with advanced epithelial ovarian, fallopian tube, or primary peritoneal cancer
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
HRD score | 2 years
  Homologous recombination deficiency score

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, M.D. Ph.D, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] da Cunha Colombo Bonadio RR, Fogace RN, Miranda VC, Diz MDPE. Homologous recombination deficiency in ovarian cancer: a review of its epidemiology and management. Clinics (Sao Paulo). 2018 Aug 20;73(suppl 1):e450s. doi: 10.6061/clinics/2018/e450s. PMID 30133561
- [Background] Bryant HE, Schultz N, Thomas HD, Parker KM, Flower D, Lopez E, Kyle S, Meuth M, Curtin NJ, Helleday T. Specific killing of BRCA2-deficient tumours with inhibitors of poly(ADP-ribose) polymerase. Nature. 2005 Apr 14;434(7035):913-7. doi: 10.1038/nature03443. PMID 15829966
- [Background] Oldenburg J, Aparicio J, Beyer J, Cohn-Cedermark G, Cullen M, Gilligan T, De Giorgi U, De Santis M, de Wit R, Fossa SD, Germa-Lluch JR, Gillessen S, Haugnes HS, Honecker F, Horwich A, Lorch A, Ondrus D, Rosti G, Stephenson AJ, Tandstad T. Personalizing, not patronizing: the case for patient autonomy by unbiased presentation of management options in stage I testicular cancer. Ann Oncol. 2015 May;26(5):833-838. doi: 10.1093/annonc/mdu514. Epub 2014 Nov 6. PMID 25378299
- [Background] Moore K, Colombo N, Scambia G, Kim BG, Oaknin A, Friedlander M, Lisyanskaya A, Floquet A, Leary A, Sonke GS, Gourley C, Banerjee S, Oza A, Gonzalez-Martin A, Aghajanian C, Bradley W, Mathews C, Liu J, Lowe ES, Bloomfield R, DiSilvestro P. Maintenance Olaparib in Patients with Newly Diagnosed Advanced Ovarian Cancer. N Engl J Med. 2018 Dec 27;379(26):2495-2505. doi: 10.1056/NEJMoa1810858. Epub 2018 Oct 21. PMID 30345884
- [Background] Lorusso D, Mouret-Reynier MA, Harter P, Cropet C, Caballero C, Wolfrum-Ristau P, Satoh T, Vergote I, Parma G, Nottrup TJ, Lebreton C, Fasching PA, Pisano C, Manso L, Bourgeois H, Runnebaum I, Zamagni C, Hardy-Bessard AC, Schnelzer A, Fabbro M, Schmalfeldt B, Berton D, Belau A, Lotz JP, Gropp-Meier M, Gladieff L, Luck HJ, Abadie-Lacourtoisie S, Pujade-Lauraine E, Ray-Coquard I. Updated progression-free survival and final overall survival with maintenance olaparib plus bevacizumab according to clinical risk in patients with newly diagnosed advanced ovarian cancer in the phase III PAOLA-1/ENGOT-ov25 trial. Int J Gynecol Cancer. 2024 Apr 1;34(4):550-558. doi: 10.1136/ijgc-2023-004995. PMID 38129136
- [Background] Ray-Coquard I, Pautier P, Pignata S, Perol D, Gonzalez-Martin A, Berger R, Fujiwara K, Vergote I, Colombo N, Maenpaa J, Selle F, Sehouli J, Lorusso D, Guerra Alia EM, Reinthaller A, Nagao S, Lefeuvre-Plesse C, Canzler U, Scambia G, Lortholary A, Marme F, Combe P, de Gregorio N, Rodrigues M, Buderath P, Dubot C, Burges A, You B, Pujade-Lauraine E, Harter P; PAOLA-1 Investigators. Olaparib plus Bevacizumab as First-Line Maintenance in Ovarian Cancer. N Engl J Med. 2019 Dec 19;381(25):2416-2428. doi: 10.1056/NEJMoa1911361. PMID 31851799